CLINICAL TRIAL: NCT01009359
Title: Open-label, Non-randomized, Multicenter Positron Emission Tomography (PET) Imaging Study to Evaluate a Single Dose of 250 MBq BAY85-8102 F-18, DPA-714 for Its Diagnostic Potential in Discriminating Patients With Probable Alzheimers Disease From Healthy Volunteers and to Evaluate the Radiation Dosimetry of a Single Dose of 150 MBq BAY858102 F-18, DPA-714 in Healthy Volunteers.
Brief Title: Evaluation of the Neuroinflammation Pattern of BAY85-8102 F-18, DPA-714 in Probable Alzheimers Disease Patients Versus Healthy Volunteers and Radiation Dosimetry of F 18, DPA-714 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer HealthCare AG
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13150; 2009-009358-26 (EudraCT Number)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Diagnostic Imaging
Keywords: Alzheimers disease; Diagnostic imaging; PET/CT diagnosis; PET tracer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: F-18 DPA-714 (BAY85-8102)
- Arm 2 (Experimental)
  Interventions: Drug: F-18 DPA-714 (BAY85-8102)
- Arm 3 (Experimental)
  Interventions: Drug: F-18 DPA-714 (BAY85-8102)

INTERVENTIONS:
Drug: F-18 DPA-714 (BAY85-8102) — Alzheimer Disease patients: Single intervenous bolus injection of 250 MBq BAY85-8102 on day one of the treatment period, PET/CT
  Arms: Arm 1
Drug: F-18 DPA-714 (BAY85-8102) — Healthy volunteers for brain imaging: Single intervenous bolus injection of 250 MBq BAY85-8102 on day one of the treatment period, PET/CT
  Arms: Arm 2
Drug: F-18 DPA-714 (BAY85-8102) — Healthy volunteers for whole body imaging: Single intervenous bolus injection of 150 MBq BAY85-8102, whole body PET/CT for evaluation of effective dose, kinetics of BAY85-8102 in blood
  Arms: Arm 3

SUMMARY:
PET (positron emission tomography) imaging with BAY85-8102 F-18, DPA-714 for investigation of neuroinflammation pattern in probable Alzheimers patients versus healthy volunteers and radiation dosimetry in healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Able to give fully informed consent in writing
* Males or females aged >/= 50 years
* No significant disease or drug use
* Absence of any sign of dementia/cognitive impairment in neuropsychological examinationsPatients for brain imaging:
* Patient and designee capable of giving fully informed consent in writing
* Patient fulfils DSM-IV and NINCDS-ADRA criteria for probable Alzheimers disease
* Patient has undergone physical and neurological examination, ECG and test of routine hematological and biochemical parameters prior to radiotracer administration Exclusion Criteria:- Pregnancy or lactation
* Current unstable medical condition (e.g. unstable angina, myocardial infarction or coronary revascularization in the preceding 12 months, cardiac failure, chronic renal failure, chronic hepatic disease, severe pulmonary disease, blood disorders, poorly controlled diabetes, chronic infection)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Discrimination of probable Alzhemimer disease patients from healthy volunteers by BAY85-81 F-18, DPA-714 brain PET imaging as evaluated by different quantification approaches | Day of Study tracer administration

SECONDARY OUTCOMES:
Discrimination of probable Alzhemimer disease patients from healthy volunteers by BAY85-81 F-18, DPA-714 brain PET imaging as evaluated by visual analysis and standard parameters(e.g. Standardized Uptake Values = SUV) | Day of Study tracer administration
Electrocardiogram (ECG) | At least once within 8 days after treatment
Blood pressure | At least 2 times within 8 days after treatment
Serum protein | At least once within 8 days after treatment
Serum creatinine | At least once within 8 days after treatment
Serum GOT (Glutamat-Oxalacetate-Transaminase) | At least once within 8 days after treatment
Adverse events collection | Continuously and for a maximum of 28 days after end of observation phase

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Turku, Finland
- Amsterdam, Netherlands